CLINICAL TRIAL: NCT04959487
Title: Food is Medicine: Randomized Trial of Medically-Tailored Food Support for Diabetes Health
Brief Title: Changing Health Through Food Support for Diabetes
Acronym: CHEFS-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Project Open Hand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK124630 (NIH); R01DK124630 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Food Insecurity
Keywords: Food security; Diabetes Mellitus; Food assistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Nutrition Assessment; Educational Status

STUDY DESIGN:
Intervention Model Description: Participants (n=440*) will be randomized to the intervention (n=220*) or control (n=220*) arms, stratified by county (San Francisco vs. Alameda County) and poor diabetes control (A1c < 9%, vs. ≥ 9%). The intervention consists of providing diabetes-tailored food support and nutritional education (two sessions of individual counseling and four session of in-group diabetes-tailored nutrition education sessions) over six months to patients with type 2 diabetes.
  *Update: Due to COVID-era challenges, NIH approved changes to the study in January 2024 including a reduced sample size (at least n=246) and reduced measures and procedures to ease participant burden (see updated Protocol/SAP Version 2, Section 7, for details).
Who Masked: Investigator
Masking Description: Single (Investigator) The investigator(s) reviewing the analyses of the data will be masked to whether participants were in the intervention or control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Control participants will receive standard of care as offered by clinical partners to all T2DM patients, including referral to nutritional counseling, T2DM support groups, and participation in local diabetes self-management programs. Control participants are also often provided referral information for locally available food support services in the region that provide diabetes-appropriate foods. At the end of follow up, the control arm will receive similar services from POH to what the intervention arm received during the intervention, regardless POH eligibility criteria (6 months of DM-tailored food support to meet 67% of their daily requirements, video recording of the 4 CHEFS-DM education classes, and access to a POH dietitian at their request).
- Food support and nutrition education (Experimental): The intervention entails two components: 1) food support that consists of weekly medically tailored meals and healthy groceries that on average covers 75% of daily energy requirements from baseline to six months and 2) diabetes-tailored nutritional education that consists of two individual counseling sessions with a Registered dietitian and four group education sessions.
  Interventions: Other: Food support; Other: Nutritional Counseling and education

INTERVENTIONS:
Other: Food support — 1. Diabetes-tailored food support. Project Open Hand will provide intervention participants six months of supplemental food support meeting on average 75% of their daily energy requirements. Food support will consist of a mix of meals tailored for T2DM, and T2DM-healthy groceries, consistent with American Diabetes Association (ADA) guidelines for diabetes healthy diets under the responsibility of a registered dietitian.
  Arms: Food support and nutrition education
Other: Nutritional Counseling and education — 2. Nutritional counseling and education: The registered dietitian will provide individual nutritional counseling two times (at baseline and month 5-6) during the intervention. In addition, group-based DM nutrition education will be conducted over four 1-hour-long sessions. The nutrition education will be conducted by a POH dietitian, and the curriculum will be consistent with published diabetes self- management education principles, utilizing effective strategies in lower wealth, lower literacy populations.
  Arms: Food support and nutrition education

SUMMARY:
This is a pragmatic randomized controlled trial (RCT) of Changing Health through Food Support for Diabetes (CHEFS-DM). This pragmatic RCT will leverage Project Open Hand's (POH) real-world programs to test the impact of a six month medically tailored food support and nutrition intervention ("CHEFS-DM") on glycemic control and other cardiometabolic outcomes, investigate the paths through which CHEFS-DM may durably improve health, and assess the economic value of the intervention to society.

DETAILED DESCRIPTION:
CHEFS-DM is a six-month intervention providing a diabetes-tailored diet meeting approximately 75% of daily energy requirements and designed based on American Diabetes Association (ADA) guidelines, together with diabetes nutritional education provided by registered dietitians. In this pragmatic RCT, investigators propose to rigorously evaluate the intervention among 440* low-income adults with Type 2 Diabetes Mellitus (T2DM) recruited from networks of safety net clinics in San Francisco and Alameda counties, California.

Participants will be randomized 1:1 to the intervention (n=220*) versus control (n=220*), using a parallel design. The study aims are as follows:

Aim 1: To determine the impact of CHEFS-DM on glycemic control and other cardiometabolic outcomes.

Aim 2: To determine the impact of CHEFS-DM on intermediate outcomes that may mediate any impact of CHEFS-DM on T2DM health.

Participant will be followed for 6 months (control arm) and 12 months (intervention arm) with structured interviews, anthropometric assessments, 24-hour dietary recalls, blood pressure measurements, blood draws, and semi structured interviews. Follow-up will be broken up into two phases. From baseline to six months, researchers will implement the CHEFS-DM intervention and follow both intervention and control arm participants (n=440*). After the end of the six-month follow-up, the intervention arm will transition to receiving standard POH services comprising 33% to 67% of daily energy requirements depending on health status, and will be followed for an additional six months, in order to assess the extent to which any health benefits are sustained at 12 months (n=220*). Hence, the control arm will be followed for six months and participate in two sets of assessments (baseline and at six months), and the intervention arm will be followed for 12 months and participate in three sets of assessments (baseline, six months, and twelve months).

*Update: Due to COVID-era challenges, NIH approved changes to the study in January 2024 including a reduced sample size (at least n=246) and reduced measures and procedures to ease participant burden (see updated SAP Version 2, Section 7, for details).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T2DM confirmed by medical or laboratory records. For T2DM, any of the following criteria will be considered (from the American Diabetes Association):

  * glycated hemoglobin (HbA1c) ≥6.5%, or
  * fasting plasma glucose of ≥126, or
  * a 2-hour plasma glucose level of 200 or higher during a 75 g oral glucose tolerance test, or
  * a random plasma glucose of 200 or higher in patients with symptoms of hyperglycemia
* Age ≥18 years.
* Screening positive for food insecurity (at least one positive answer) in the previous 6 months assessed using the 6-item version of the US Household Food Security Survey Module (US Department of Agriculture), or has household income <200% of the federal poverty level.
* English or Spanish language fluency.
* Adequate cognitive and hearing capacity to consent and complete study measures.
* Reside in Alameda County or San Francisco County.

Exclusion Criteria:

* Type-1 diabetes mellitus
* Individuals with disorders known to affect the accuracy of the HbA1c measure (e.g., end stage renal disease and individuals with known hemoglobinopathies).
* Inability to attend the educational workshops.
* Inability to schedule baseline assessments and/or blood draw after repeated requests.
* Pregnant individuals, or individuals planning to get pregnant within 6 months, or are lactating, or are postpartum less than 6 months.
* Current POH clients, past POH clients who stopped services less than 6 months prior, or past or present participants in other POH medically tailored meals studies.
* Does not have access to food storage, including a refrigerator and freezer to safely keep food.
* Does not have access to facilities to reheat and prepare meals using Project Open Hand food.
* Anticipates moving out of study area of Alameda and San Francisco Counties in the next 6 months.
* Receives more than 1 meal per day from a free food support resource or agency.
* Allergic to or will not eat eggs, soy, wheat, nuts, seeds or seed oils, or other foods commonly included among ingredients in POH meals.
* Allergic to dairy products, or unable to tolerate any dairy products including milk, yogurt and cheese.
* Individual does not eat any or all of POH's meat meal options and will not eat the vegetarian POH meal option.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c from baseline to six months by study arm | Baseline and six months
  Change HbA1c levels (%) from baseline to six months by study arms.
Change in food insecurity severity from baseline to six months by study arm | Baseline and six months
  The US adult food security survey module from the US Department of Agriculture (USDA) will be used to assess the change in the food security scores from baseline to six months. The score ranges from 0 to 10. Higher score indicates higher severity of food insecurity

SECONDARY OUTCOMES:
Change in the proportion of participants with low and very low food security | Baseline and six months
  Low and very low food security will be defined as 3 or more items answered affirmatively in the USDA's US adult food security survey module. Change in proportion of participants with low or very low food security, from baseline to six months by intervention arms will be reported.
Change in proportion of participants with glucose control by study arm. | Baseline and six months
  Glucose control will be defined as HbA1c lower than 9%. The change from baseline to six months, in the proportion of participants with glucose control will be reported.
Change in systolic and diastolic blood pressure from baseline to six months | Baseline and 6 months
  Changes in the average of three repeated measurements of systolic and diastolic blood pressure (mm Hg) from baseline to six months by study arm.
Change in medication adherence from baseline to six months by study arm | Baseline and six months
  A single-item Rating Visual Analogue Scale will be used to evaluate diabetes medication adherence. Using the scale, participants self-report the adherence of medication ranging from 0% to 100%. The changes in diabetes medication adherence (percentage) from baseline to six months by study arms will be reported.
Acute health care utilization from baseline to six month by study arm | Baseline and six months
  Proportion of participants that used emergency health care (Emergency department or urgent care) during the 6 months of the study by study arm will be reported.
Hospital admissions from baseline to six months by study arm | Baseline to six months
  Proportion of participants who were hospitalized at least once from baseline to six months of the study by study arms will be reported.
Missed outpatient visits from baseline to six months by study arm | Baseline to six months
  Proportion of participants that missed at least one outpatient visits from baseline to six months by study arms will be reported.
Change in health-related quality of life scores from baseline to six months by study arm | Baseline and six months
  The quality of life will be measured using the standardized 12-item short form health survey (SF-12v2). The SF-12v2 provides a summary score for physical and mental health. The transformed T score has a mean=50 and Standard Deviation=10, in which higher values means better health. The change in SF-12 T scores from baseline to six months by study arm will be reported.
Change in body mass index (BMI) from baseline to six months by study arm | Baseline and six months
  The average of three repeated measurements of weight and height will be obtained at baseline and at six months. The BMI will be calculated (weight (kg)/ (height (m)^2). Changes in in BMI values (kg/ m^2) from baseline to six months by study arm will be reported.
Change in healthy eating index score 2015 (HEI-2015) from baseline to six months by study arm. | Baseline and six months
  Dietary information using an automated self- administered 24-hour dietary recall instrument from the National Cancer Institute's (ASA24) will be collected. The HEI-2015 is a measure of diet quality which evaluates how well the food consumed aligns with the Dietary guidelines for American population. The HEI-2015 score ranges from 0-100 in which a higher score indicates better diet quality. The adequacy component of the HEI ranges from 0-60 and the moderation component ranges from 0-40 (both with higher score indicating better diet quality). Changes in the adequacy and moderation HEI-2015 score from baseline to six months by study arm will be reported.
Change in depressive symptoms from baseline to six months by study arm | Baseline and six months
  The 9-item Patient Health Questionnaire (PHQ-9) will be used to evaluate depressive symptoms. The PHQ-9 score ranges from 0 to 27, with higher scores indicating higher levels of depression. The change in PHQ-9 scores from baseline to six months by study arm will be reported.
Change in diabetes distress scale from baseline to six months by study arm | Baseline and six months
  The diabetes distress scale (DDS) has 17 items measuring frustration, anger, and discouragement associated with managing complex diabetes health-care directives. The DDS score ranges from 1 to 6, with higher scores indicating higher levels of distress. The change in diabetes distress scores from baseline to six months by study arms will be reported.
Change in diabetes self-efficacy from baseline to six months by study arm | Baseline and six months
  The 8-item Perceived Diabetes Self-Management (PDSM) scale will be used to assess confidence in one's ability to manage numerous self-care behaviors, including diet, and management of glucose. The PDSM scores ranges from 8 to 40, with higher scores indicating more confidence in self-managing their diabetes. The changes in the PDSM scores from baseline to six months by study arm will be reported.

OTHER OUTCOMES:
Durability of HbA1c values from six months to twelve months in the intervention arm. | Six and twelve months
  To evaluate durability of the HbA1c after the intervention ended, the change in HbA1c levels (%) from six months to twelve months in the intervention group will be reported.
Durability in scores of food security from six to twelve months in the intervention arm. | Six and twelve months
  To evaluate durability of food security after the intervention ended, the change in food insecurity scores from six months to twelve months in the intervention group will be reported. The US adult food security survey module from the USDA will be used. The score ranges from 0 to 10. Higher score indicates higher severity of food insecurity.

CONTACTS AND LOCATIONS:
Overall Officials: Kartika Palar, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Project Open Hand, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palar K, Napoles T, Hufstedler LL, Seligman H, Hecht FM, Madsen K, Ryle M, Pitchford S, Frongillo EA, Weiser SD. Comprehensive and Medically Appropriate Food Support Is Associated with Improved HIV and Diabetes Health. J Urban Health. 2017 Feb;94(1):87-99. doi: 10.1007/s11524-016-0129-7. PMID 28097614
- [Background] Seligman HK, Lyles C, Marshall MB, Prendergast K, Smith MC, Headings A, Bradshaw G, Rosenmoss S, Waxman E. A Pilot Food Bank Intervention Featuring Diabetes-Appropriate Food Improved Glycemic Control Among Clients In Three States. Health Aff (Millwood). 2015 Nov;34(11):1956-63. doi: 10.1377/hlthaff.2015.0641. PMID 26526255
- [Background] Seligman HK, Schillinger D. Hunger and socioeconomic disparities in chronic disease. N Engl J Med. 2010 Jul 1;363(1):6-9. doi: 10.1056/NEJMp1000072. No abstract available. PMID 20592297
- [Background] Gurvey J, Rand K, Daugherty S, Dinger C, Schmeling J, Laverty N. Examining health care costs among MANNA clients and a comparison group. J Prim Care Community Health. 2013 Oct;4(4):311-7. doi: 10.1177/2150131913490737. Epub 2013 Jun 3. PMID 23799677
- [Background] Berkowitz SA, Terranova J, Hill C, Ajayi T, Linsky T, Tishler LW, DeWalt DA. Meal Delivery Programs Reduce The Use Of Costly Health Care In Dually Eligible Medicare And Medicaid Beneficiaries. Health Aff (Millwood). 2018 Apr;37(4):535-542. doi: 10.1377/hlthaff.2017.0999. PMID 29608345
- [Background] Berkowitz SA, Terranova J, Randall L, Cranston K, Waters DB, Hsu J. Association Between Receipt of a Medically Tailored Meal Program and Health Care Use. JAMA Intern Med. 2019 Jun 1;179(6):786-793. doi: 10.1001/jamainternmed.2019.0198. PMID 31009050
- [Background] Seligman HK, Jacobs EA, Lopez A, Tschann J, Fernandez A. Food insecurity and glycemic control among low-income patients with type 2 diabetes. Diabetes Care. 2012 Feb;35(2):233-8. doi: 10.2337/dc11-1627. Epub 2011 Dec 30. PMID 22210570
- [Background] Seligman HK, Jacobs EA, Lopez A, Sarkar U, Tschann J, Fernandez A. Food insecurity and hypoglycemia among safety net patients with diabetes. Arch Intern Med. 2011 Jul 11;171(13):1204-6. doi: 10.1001/archinternmed.2011.287. No abstract available. PMID 21747017
- [Background] Marpadga S, Fernandez A, Leung J, Tang A, Seligman H, Murphy EJ. Challenges and Successes with Food Resource Referrals for Food-Insecure Patients with Diabetes. Perm J. 2019;23:18-097. doi: 10.7812/TPP/18-097. PMID 30939269

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT04959487/Prot_SAP_001.pdf